CLINICAL TRIAL: NCT03529344
Title: A 6-week Pilot Study to Investigate the Effects of Protein Hydrolysate From Blue Whiting on Glucose Regulation, Inflammation and Serum Lipids in Elderly Nursing Home Residents From Western Norway
Brief Title: A Study on the Effects on Glucose Regulation, Inflammation and Serum Lipids After Fish Protein Supplementation in Elderly (GRIPE)
Acronym: GRIPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bergen (Other)
Responsible Party: Principal Investigator, Oddrun Anita Gudbrandsen, Principal Investigator, University of Bergen
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2015/75
Record Dates: First submitted 2018-05-07; First posted 2018-05-18 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2022-01

CONDITIONS: Muscle Weakness; Muscle Loss; Blood Sugar; High; Inflammation; Aging
MeSH Terms: conditions — Muscle Weakness; Muscular Atrophy; Hyperglycemia; Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blue whiting protein hydrolysate (Active Comparator): Dietary Supplement: Blue whiting protein hydrolysate 6g protein per day for 6wk
  Interventions: Dietary Supplement: Blue whiting protein hydrolysate
- Placebo Comparator: Control (Placebo Comparator): Control group will receive non-caloric juice without protein supplementation
  Interventions: Dietary Supplement: Placebo Comparator: Control

INTERVENTIONS:
Dietary Supplement: Blue whiting protein hydrolysate — Dietary Supplement: Blue whiting protein hydrolysate 6g protein per day for 6wk
  Arms: Blue whiting protein hydrolysate
Dietary Supplement: Placebo Comparator: Control — Control group will receive non-caloric juice without protein supplementation
  Arms: Placebo Comparator: Control

SUMMARY:
The elderly population have and increased risk of loss of both muscle mass and function and is therefore recommended a higher protein intake than the healthy adult population. These age-related changes in muscle function may be explained by chronic low-grade inflammation and insulin resistance. Despite the recommendation of a higher protein intake, little is known about how different protein sources may affect the metabolic health in this population. Analysis of amino acid composition show that fish can be a good protein source for humans. Many fish species are today used as feed ingredients, rather than a protein source for humans. A few studies conducted in humans and rats show that proteins from fish may improve glucose tolerance, reduce inflammation and improve lipid metabolism, indicating that proteins from fish may not only serve as a valuable nutrient but could also hold specific health promoting properties.

The present study will investigate the effects of a protein hydrolysate from blue whiting, a fish species normally used to produce fish meal for aquaculture industry, on glucose homeostasis, inflammation and serum lipids in elderly nursing home residents.

DETAILED DESCRIPTION:
Participants receive 6g per day of protein hydrolysate from blue whiting as protein powder mixed with a non-caloric juice for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* >60 years
* both genders
* nursing home resident

Exclusion Criteria:

* life expectancy < 6 months
* severe cognitive impairment
* allergies towards fish, milk, egg
* weight loss >5% last 3 months

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Participant compliance | 6 weeks
  Investigate the participant compliance based daily registrations by nursing home staff
Participant dropout rate | 6 weeks
  Number of participants that completed the intervention period

SECONDARY OUTCOMES:
Glucose regulation | 6 weeks
  Glucose concentration will be measured in fasting serum
Insulin | 6 weeks
  Insulin will be measured in fasting serum/plasma
C-reactive protein in serum | 6 weeks
  C-reactive protein (a marker of inflammation) will be analysed in fasting serum
Interleukin-6 in serum | 6 weeks
  Interleukin-6 (a marker of inflammation) will be analysed in fasting serum
Monocyte chemoattractant protein-1 in serum | 6 weeks
  Monocyte chemoattractant protein-1 (a marker of inflammation) will be analysed in fasting serum

CONTACTS AND LOCATIONS:
Overall Officials: Oddrun A Gudbrandsen, PhD, Principal Investigator — University of Bergen

REFERENCES:
- [Result] Drotningsvik A, Oterhals A, Flesland O, Nygard O, Gudbrandsen OA. Fish protein supplementation in older nursing home residents: a randomised, double-blind, pilot study. Pilot Feasibility Stud. 2019 Feb 26;5:35. doi: 10.1186/s40814-019-0421-x. eCollection 2019. PMID 30858985